CLINICAL TRIAL: NCT01344954
Title: Single Intravenous Administration of TB-402 for the Prophylaxis of Venous Thromboembolic Events (VTE) After Total Hip Replacement Surgery: A Phase 2b, Multicentre, Randomised, Active-Controlled, Double Blind, Double Dummy, Parallel Group Study
Brief Title: Single IV Administration of TB-402 for Prophylaxis of Venous Thromboembolic Events (VTE) After Total Hip Replacement Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Collaborators: BioInvent International AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TB-402-006
Record Dates: First submitted 2011-03-18; First posted 2011-04-29 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Prophylaxis of Venous Thromboembolic Events
MeSH Terms: interventions — TB 402; Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 25mg TB-402 (Experimental)
  Interventions: Drug: TB-402
- 50mg TB-402 (Experimental)
  Interventions: Drug: TB-402
- 10mg QD Rivaroxaban (Active Comparator)
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: TB-402 — Administered intravenously over 10 minutes
  Arms: 25mg TB-402
Drug: Rivaroxaban — Administered orally as a capsule once a day for 35 days
  Other Names: Xarelto
  Arms: 10mg QD Rivaroxaban
Drug: TB-402 — Administered intravenously over 10 minutes
  Arms: 50mg TB-402

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of two doses of TB-402 administered as a single intravenous infusion for the prevention of VTE in subjects undergoing total hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years.
2. Written informed consent.
3. Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

1. Pregnancy at the time of screening.
2. Indication for anticoagulation other than post-operative thromboprophylaxis.
3. Active bleeding or high risk of bleeding.
4. Anticipated continued use of neuraxial catheter after surgery.
5. Clinical laboratory findings at screening of thrombocytopenia or prolonged aPTT or PT.
6. Uncontrolled hypertension.
7. Impaired liver function (transaminase >3 X ULN) or history of hepatic insufficiency.
8. Creatinine clearance <30 mL/min.
9. Antiplatelet agents other than low dose aspirin (< 200mg).
10. The use of intermittent pneumatic compression.
11. Known hypersensitivity to contrast media or rivaroxaban.
12. Known drug or alcohol abuse.
13. Active malignant disease or current cytostatic treatment.
14. Stroke within the previous month.
15. Participation in an investigational drug study within the past 30 days or previous participation in this study.
16. Any condition that in the opinion of the investigator would put the subject at increased risk from participating in the study or expected inability to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Composite of asymptomatic DVT as detected by bilateral venography and symptomatic VTE, i.e. DVT or fatal or non-fatal PE | Randomisation to post-operative day 35

SECONDARY OUTCOMES:
Incidents of major VTE | Randomisation to Post-Operative day 35
Incidents of total DVT | Randomisation to Post-Operative day 35
Incidents of proximal/distal DVT | Randomisation to Post-Operative day 35
Incidents of pulmonary embolism | Randomisation to Post-Operative day 35
Incidents of VTE-related death | Randomisation to Post-Operative day 35
Incidents of Major VTE | Randomisation to Post-Operative day 70

CONTACTS AND LOCATIONS:
Locations (36):
- Austria (4):
  - KRANKENHAUS DES BARMHER.SCHW.Linz, Linz
  - AKH Wien, Vienna
  - Orthopädisches Spital Speising, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- ZNA Antwerpen Locatie Middelheim, Antwerp, Belgium
- Bulgaria (5):
  - SHAT of orthopedics, traumatology and surgery "Sv. Pantaleimon " - Pleven Department of Orthopaedics and Traumatology, Pleven
  - Department of Orthopedics, UMHAT "Sv. Georgi", Plovdiv
  - MHAT Rousse, Department of Orthopaedics, Rousse
  - UMHAT "St Anna" AD,Clinic of Orthopaedics and Traumatology, Sofia
  - UMHAT 'Tsaritsa Joanna', Sofia
- Hungary (3):
  - Pándy Kálmán Kórház, Gyula
  - Bács-Kiskun Megyei Önkormányzat Kórháza, Szegedi Tudományegyetem Általános Orvostudományi Karháza, Kecskemét
  - Tolna Megyei Önkormányzat Balassa János Kórháza, Szekszárd
- Latvia (4):
  - Traumatology and Orthopedics Clinic "Adazi", LTD, Ādaži
  - Ltd "Liepajas regionala slimnica", Liepāja
  - Riga 2nd Hospital, Riga
  - Ltd "Vidzemes slimnica", Valmiera
- Diaconessenhuis Leiden, Leiden, Netherlands
- Poland (5):
  - Klinika Orthopedii I Traumatologii, Bialystok
  - Wojewódzkie Centrum Ortopedii i Rehabilitacji Narządu Ruchu im. dr Z. Radlińskiego w Łodzi, Lodz
  - NZOZ Szpital w Puszczykowie, Puszczykowo
  - Klinika Ortopedii, WIM, Warsaw
  - Medical University of warsaw, Dept of Orthopaedics, Warsaw
- Russia (7):
  - Municipal Healthcare Institution "City Clinical Hospital No. 3", Chelabinsk
  - Municipal Healthcare Medical Institution "City Clinical Hospital No. 4", Orenburg
  - Federal State Healthcare Institution: Clinical Hospital #122 named after L.G. Sokolov under the Federal Medical-Biological Agency of Russia, Saint Petersburg
  - Saint Petersburg State Healthcare Institution "City Aleksandrovskaya Hospital", Saint Petersburg
  - Saint Petersburg State Healthcare Institution "Municipal Multi-Speciality Hospital No. 2", Saint Petersburg
  - State Healthcare Institution "Samara Regional Clinical Hospital n.a. M.I. Kalinin", Samara
  - Municipal Healthcare Institution "Clinical Hospital of Emergency Care n.a. N.V. Soloviov", Yaroslavl
- Ukraine (6):
  - Public Entity "Regional Hospital - Center of Emergency Medical Care and Disaster Medicine" of Cherkasy Regional Council, Department of orthopedy and traumatology, Cherkassy
  - Ivano-Frankіvsk Regional Clinical Hospital MoH Ukraine, Department of ortopedics and traumatology. Department of traumatology, ortopedics and military/emergency surgery of Ivano-Frankіvsk National Medical University, Ivano-Frankivsk
  - SE "Sytenko Institute of Spine and Joint Pathology, AMS Ukraine", department of orthopedic arthrology and endoprosthesis replacement, Kharkiv
  - Public Entity of Kyiv Regional council "Kyiv Regional Clinical Hospital", Ortopedy and traumatology center of Public Entity of Kyiv Regional council "Kyiv Regional Clinical Hospital", Kyiv
  - Public Establishment "Odessa Regional Clinical Hospital", Department of Orthopedics and Traumatology., Odesa
  - Public Establishment 'City Hospital #9', orthopedy and traumatology department, Sevastopol